CLINICAL TRIAL: NCT03923556
Title: A Double-blind, Randomized, Parallel Study to Compare the Efficacy of Sugammadex Versus Neostigmine for Reversal of Neuromuscular Blockade at the End of Kidney Transplantation Surgery in Patients With Severe Kidney Dysfunction
Brief Title: Sugammadex Versus Neostigmine for Reversal of Neuromuscular Blockade at the End of Kidney Transplantation Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 18-2707
Record Dates: First submitted 2019-03-28; First posted 2019-04-22 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Kidney Transplant; Complications; Postoperative Residual Curarization; Postoperative Residual Weakness
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sugammadex (Experimental): Sugammadex
  Interventions: Drug: Sugammadex
- Neostigmine (Active Comparator): Neostigmine
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — Administration of Sugammadex intravenously at a dose appropriate for the reversal of neuromuscular blockade (usually 2-4 mg/kg) at the end of the surgery before tracheal extubation
  Arms: Sugammadex
Drug: Neostigmine — Administration of Neostigmine intravenously at a dose appropriate for the reversal of neuromuscular blockade (usually 0.03-0.07 mg/kg) at the end of the surgery before tracheal extubation
  Arms: Neostigmine

SUMMARY:
The purpose of this study is to compare two medications that reverse muscle paralysis at the end of kidney transplant surgery with the goal of reducing residual muscle weakness and insufficient respiratory function after surgery.

DETAILED DESCRIPTION:
This is a prospective randomized double-blind single center study on patients with severe kidney failure undergoing kidney transplantation surgery. Patients will have their muscles paralyzed during general anesthesia for surgery. At the end of surgery, muscle paralysis will be reversed with either neostigmine (control group) or sugammadex (intervention group). Residual muscle weakness and respiratory function will be monitored after surgery with a quantitative train-of-four (qTOF) monitor and a noninvasive continuous ventilation monitor. The investigators hypothesize that patients receiving sugammadex will have less residual muscle weakness and better respiratory function than patients receiving neostigmine. Respiratory and kidney function parameters and any adverse events will be collected during the hospital stay. Patients will contacted for a study follow up around 2 weeks after their surgery.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years or older
* Diagnosed with severe kidney dysfunction (defined by plasma creatinine clearance <30 mL/min)
* Planning on kidney transplantation surgery at the University of Colorado Hospital.

Exclusion Criteria:

* Patients unable to sign the informed consent
* Pregnant women
* Body Mass Index (BMI) > 40 kg/m2
* Pre-existing oxygen or ventilatory dependency (24h use of oxygen or other noninvasive or invasive ventilatory support)
* Patients with any pulmonary, neuromuscular or other disease that severely limits their respiratory functional status (e.g. unable to achieve 4 Metabolic Equivalent of Tasks, METs, such as climbing up 1 flight of stairs)
* Presence of any contraindication for any of the study-related medications or interventions.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Fernandez-Bustamante, M.D., Ph.D., Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugammadex | Neostigmine
Started | 42 | 42
Completed (2 participants in each group lacked sufficient information for primary outcome assessment) | 42 (received assigned protocol) | 42 (received assigned protocol)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Neostigmine | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [38 to 56] | 53 [37 to 64] | 50 [37 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 21 | 32
  Male | 31 | 21 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 30 | 26 | 56
  Race/Ethnicity: Hispanic or Latino | 9 | 7 | 16
  Race/Ethnicity: Other | 3 | 9 | 12
Preoperative hemodialysis [Count of Participants; unit: Participants] | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Hypoventilation in Post-anesthesia Care Unit (PACU)
Description: Presence of one or more episodes of hypoventilation in PACU, adjusted to qTOF and other confounders
Time Frame: Within up to 3 hours after the end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 40 | 40
Participants | 22 | 23

2. Secondary Outcome: Number of Patients With Presence of qTOF <0.9 in PACU
Description: Incidence of qTOF <0.9 in PACU
Time Frame: Within up to 3 hours after the end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 42 | 42
Participants | 13 | 25

3. Secondary Outcome: Number of Participants With Kidney Graft Dysfunction
Description: Predefined kidney graft negative outcomes including: postoperative increasing ClCr, reduced daily urine output, need for dialysis postoperatively, and/or diagnosis of delayed graft function or kidney graft rejection.
Time Frame: Within up to 3 postoperative days and at 14 +/- 3 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 42 | 42
Participants | 2 | 4

4. Secondary Outcome: Rate of Adverse Events Related to NMBR Medications
Description: Adverse events related to NMBR medications, including hypersensitivity and any other adverse events
Time Frame: Within up to 3 postoperative days
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 42 | 42
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: First 2 postoperative weeks
Description: Following definitions and processes described in protocol.
Arm/Group | Sugammadex | Neostigmine
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 4/42 | 4/42
Other Adverse Events (participants affected / at risk) | 2/42 | 1/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sugammadex (N=42) | Neostigmine (N=42)
Postoperative ureteral leak (Renal and urinary disorders) | 1 | 0
Cerebrovascular accident (Vascular disorders) | 0 | 1
Reoperation for bleeding (Vascular disorders) | 1 | 1
Kidney graft dysfunction (Renal and urinary disorders) | 2 | 1
Opioid-induced respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sugammadex (N=42) | Neostigmine (N=42)
Respiratory symptoms requiring oxygen supplementation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT03923556/Prot_SAP_000.pdf